CLINICAL TRIAL: NCT03536364
Title: Effect of Food Order on Postprandial Glucose Excursions in Pre-Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1612017822
Record Dates: First submitted 2018-03-23; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Obesity; Pre-Diabetes
MeSH Terms: conditions — Obesity; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prediabetes (Experimental): manipulation of food order during a meal on postprandial in subjects with prediabetes
  Interventions: Behavioral: Food Order; Behavioral: Carbohydrate Last; Behavioral: Vegetables first

INTERVENTIONS:
Behavioral: Food Order — carbohydrate (ciabatta bread ) first, followed 10 minutes later by protein (grilled chicken) and vegetables
  Other Names: Carbohydrate First
Behavioral: Carbohydrate Last — protein and vegetables first, followed 10 minutes later by carbohydrate
Behavioral: Vegetables first — vegetables first, followed 10 mins later by protein and carbohydrate.

SUMMARY:
The natural history of type 2 diabetes commonly follows a pattern of postprandial dysregulation followed by fasting hyperglycemia leading to overt type 2 diabetes. Approximately 38% of the US adult population is estimated to have pre-diabetes. In a previous study of 16 overweight/obese patients with metformin treated type 2 diabetes, using a typical Western meal, investigators demonstrated that a food order in which protein and vegetables are consumed first, before carbohydrate, results in significant lowering of incremental glucose peaks compared to the reverse order. In the present study, investigators seek to expand on the previous findings to gain further insight into the impact of food order in individuals with pre-diabetes, using a meal with different macronutrient composition, in the setting of three meal patterns. The study is designed to be a simple, practical intervention that may have very significant clinical implications for prevention of diabetes in a large population at increased metabolic risk.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 30-65 years of age
2. BMI 25-40kg/m2
3. HbA1c 5.7%-6.4%
4. Willing to comply with study requirements
5. Provide written informed consent

Exclusion Criteria:

1. Known diagnosis of diabetes / taking any medication for treatment of diabetes
2. History of previous bariatric surgery
3. History of chronic liver or renal disease
4. Current treatment with systemic corticosteroids
5. Pregnant women
6. History of allergy to any component of the test meal

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Effect of food order on postprandial glucose excursions as measured by incremental glucose peaks (mg/dl) in the setting of 3 commonly followed meal patterns in overweight/obese patients with pre-diabetes | 30, 60, 90, 120, 150 and 180 mins
Effect of food order on postprandial glucose excursions as measured by post prandial glucose levels (mg/dl) in the setting of 3 commonly followed meal patterns in overweight/obese patients with pre-diabetes | 30, 60, 90, 120, 150 and 180 mins
Effect of food order on postprandial glucose excursions as measured by incremental area under the curve (iAUC) for glucose ((mg/dl)*180) in the setting of 3 commonly followed meal patterns in overweight/obese patients with pre-diabetes | 0-180 min

SECONDARY OUTCOMES:
Effect of food order on postprandial insulin levels (microIU/ml) in the setting of 3 commonly followed meal patterns in overweight/obese patients with pre-diabetes | 30, 60, 90, 120, 150 and 180 mins
Effect of food order on postprandial insulin incremental area ((microIU/ml)*180min) under the curve in the setting of 3 commonly followed meal patterns in overweight/obese patients with pre-diabetes | 0-180 mins
Effect of food order on satiety as measured by a visual analog scale (cm) in the setting of 3 commonly followed meal patterns in overweight/obese patients with pre-diabetes | 0,60,120, and 180 mins

CONTACTS AND LOCATIONS:
Overall Officials: Alpana P Shukla, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Comprehensive Weight Control Center, New York, New York, United States